CLINICAL TRIAL: NCT01825148
Title: Clinical Proof-of-principle of the Determination of the Beta Cell Mass in Vivo by SPECT Imaging With the 111-In-labeled GLP-1 Analogue DTPA(Diethylenetriamine Pentaacetic Acid)-[K40]-Exendin 4
Brief Title: GLP-1 Receptor Targeting in Diabetic and Healthy Individuals
Acronym: GLP-1-CPOP
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Martin Gotthardt, Prof. Dr., Radboud University Medical Center
Other Study IDs: RUNMC-EX-BCM-2012; 2012-000619-10 (EudraCT Number)
Record Dates: First submitted 2013-03-18; First posted 2013-04-05 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Type 1 Diabetes: patients with long standing T1D
  Interventions: Other: radiolabeled Exendin
- Healthy volunteer: healthy volunteers with normal glucose tolerance
  Interventions: Other: radiolabeled Exendin

INTERVENTIONS:
Other: radiolabeled Exendin

SUMMARY:
The purpose of the study is to determine whether there are differences in pancreatic uptake of the radiotracer between healthy individuals and patients with type 1 diabetes. If T1D patients have a markedly reduced uptake, the compound may be suitable for estimation of pancreatic beta cell mass, i.e. the cells in the pancreas that produce insulin.

ELIGIBILITY:
Inclusion Criteria:

* type 1 Diabetes

Exclusion Criteria:

* breast feeding
* pregnant

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Type 1 Diabetes patients and healthy volunteers responding to advertisment
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
pancreatic uptake of radiolabeled Exendin | 7 days
  uptake will be given as counts per MBq injected activity as determined by calibrated SPECT/CT scanner with attenuation correction.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Brom M, Woliner-van der Weg W, Joosten L, Frielink C, Bouckenooghe T, Rijken P, Andralojc K, Goke BJ, de Jong M, Eizirik DL, Behe M, Lahoutte T, Oyen WJ, Tack CJ, Janssen M, Boerman OC, Gotthardt M. Non-invasive quantification of the beta cell mass by SPECT with (1)(1)(1)In-labelled exendin. Diabetologia. 2014 May;57(5):950-9. doi: 10.1007/s00125-014-3166-3. Epub 2014 Feb 1. PMID 24488022